CLINICAL TRIAL: NCT05539092
Title: Faculty of Nursing- Critical Care and Emergency Nursing Department
Brief Title: The Effect of Changing Angle of Bed on Pain Severity and Vascular Complications Among Cardiac Catheterization Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, sara sobh mohamed ramadan ellawindy, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ref.no.p 0.0237
Record Dates: First submitted 2022-08-25; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Catheterization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): the researcher will change angle of bed from 15° to 45°. The severity of pain will be assessed for five times starting immediately after sheath removal. Vascular complications monitoring scales will be assessed I for five times starting immediately after sheath removal.
  Interventions: Other: changing angle of bed
- control group (No Intervention): positioning the patients in supine for 6 hours and the affected leg was straight and immobilized. The severity of pain will be assessed for five times starting immediately after sheath removal. Vascular complications monitoring scales will be assessed I for five times starting immediately after sheath removal.

INTERVENTIONS:
Other: changing angle of bed — Before the cardiac catheterization procedure: patients' demographic characteristics and health relevant data will be collected on the first day of admission. the researcher will change angle of bed from 15° to 45°.
  Arms: intervention group

SUMMARY:
Care of CVD patients in Egypt is very complex and sensitive because of the high incidence and high mortality rate. In 2019, approximately 18.6 million deaths were attributed to CVD globally. As a consequence, cardiac catheterization remains the criterion standard for evaluation of CAD.

DETAILED DESCRIPTION:
This study will be conducted in three phases; preparation, implementation, and evaluation.

1. Preparation phase

   * Ethical approval will be obtained from the Research Ethics Committee (REC) of the Faculty of Nursing - Mansoura University.
   * Content validity of the developed tool will be reviewed by a jury of five experts in the study field and the suggestions of the jury members will be considered.
   * The reliability of this tool will be assessed also by using Cronbach's Alpha Test.
2. Implementation phase

   * An initial assessment will be carried out for all patients to confirm that they are free from the exclusion criteria.
   * Patients will be assigned into two groups: intervention group and control group, 41 patients for each group.
   * Before the cardiac catheterization procedure: patients' demographic characteristics and health relevant data will be collected on the first day of admission using part I and part II of tool I.
   * In both groups after cardiac catheterization procedure: the sheath will be removed immediately by the nurse.
   * In the control group: positioning the patients in supine for 6 hours and the affected leg was straight and immobilized.
   * In the intervention group: the researcher will change angle of bed from 15° to 45°.
   * The severity of pain will be assessed by using part III of tool I for five times starting immediately after sheath removal.
   * Vascular complications monitoring scales will be assessed by using tool III for five times starting immediately after sheath removal.
3. Evaluation phase This phase aims to investigate the effect of changing angle of bed on pain severity and vascular complications for both groups.

ELIGIBILITY:
Inclusion Criteria:

Adult patient ≥ 18 years old of both sexes.

* Conscious patients admitted to the CCU after diagnostic or therapeutic cardiac catheterization.
* Patients who will have femoral artery catheterization.
* Patients who will have normal prothrombin time and partial thromboplastin time.

Exclusion Criteria:

* Patients who have previous surgery in the iliac or femoral artery.

  * Patients who have chronic back pain.
  * Patients who have an active bleed¬ing, hematoma and ecchymosis from insertion site prior to the sheath withdrawal.
  * Patient who take anti-coagulant drugs and analgesic therapy within the previous 24 hours before the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
changing pain severity according to the numerical pain scale | 6 hours
  Patients who receive changing angle of bed after cardiac catheterization will have less pain severity according to the numerical pain scale than those who will receive hospital routine care.

SECONDARY OUTCOMES:
reduction of vascular complications according to the vascular complications monitoring scales | 6 hours
  The vascular complications will be decreased after changing angle of bed among cardiac catheterization patients according to the vascular complications monitoring scales